CLINICAL TRIAL: NCT06971549
Title: Accelerated iTBS for Depression: Monitoring Brain Hemodynamics With Simultaneous iTBS/fNIRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Georg Kranz, Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSEARS20230705001-01
Record Dates: First submitted 2025-04-27; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Depression
Keywords: Theta-Burst stimulation (iTBS); Functional near-infrared spectroscopy (fNIRS); Concurrent TMS/fNIRS; Prefrontal hemodynamic response
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerating TMS teatment (Experimental): One depressed patient will be included in this study, which lasts for 5 consecutive days. During these 5 days, the participant will receive accelerated TMS treatment based on SAINT protocol, simultaneously monitored by concurrent TMS/fNIRS.
  Interventions: Other: Accelerated iTBS

INTERVENTIONS:
Other: Accelerated iTBS — Fifty iTBS sessions (1,800 pulses per session, 50-minute intersession interval) will be delivered as 10 daily sessions over 5 consecutive days at 90% resting motor threshold.

SUMMARY:
This study will investigate the cortical hemodynamic response variability of an accelerated form of TBS stimulation over left dorsolateral prefrontal cortex (DLPFC) using a concurrent TBS/fNIRS setup. The accelerating TMS protocol that will be used in this study is similar to the Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT), i.e., fifty iTBS sessions (1,800 pulses per session, 50-minute intersession interval) will be delivered as 10 daily sessions over 5 consecutive days at 90% resting motor threshold. The investigators will recruit a depressed patient and conduct a concurrent iTBS/fNIRS protocol for each iTBS session. Moreover, the depression symptoms of the patient will be assessed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 65;
* a clinical diagnosis of current nonpsychotic major depressive disorder by an experienced psychiatrist according to DSM-IV;
* no or stable (≥2 weeks) psychopharmacological medication;
* have not responded to at least one antidepressant medication;
* have not received any TMS treatment;
* and have a 17-item HAMD score ≥ 20.

Exclusion Criteria:

* severe internal diseases;
* neurological disorders or a history of severe head injuries;
* having suicidal ideation;
* pregnancy;
* common MRI, fNIRS and TMS exclusion criteria, such as a history of brain surgery, head injury, cardiac pacemaker, deep brain stimulation, intracranial metallic particles, history of seizures
* antiepileptics and benzodiazepines corresponding to a dose of >1 mg lorazepam/d.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Oxygenated and deoxygenated hemoglobin (HbO and HbR) change compared to baseline | Before, during and immediately after the intervention
  iTBS-induced HbO and HbR change in the DLPFC before, during and after stimulation
Hamilton Depression Rating Scale (HAM-D) | through study completion, an average of 5 days
  The Hamilton Depression Rating Scale, 17 item (HAM-D-17) is a simple, clinician-administered tool used to assess symptoms of depression experienced by a patient in the past week. The values of HAM-D-17 range from 0 to 52, and higher socres mean more severe symptoms.

SECONDARY OUTCOMES:
Montgomery-Asberg depression rating scale (MADRS) | through study completion, an average of 5 days
  The Montgomery-Åsberg Depression Rating Scale is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
Patient Health Questionnaire-9 (PHQ-9) | daily for 5 days
  Patient Health Questionnaire-9 (PHQ-9) is a 9-question instrument to screen for depression. Each item yields a score of 0 to 3; the overall score thus ranges from 0 to 27. Higher PHQ-9 score indicates more severe depression.
Verbal Analogue Scale (VAS) fatigue and pain level | immediately after the intervention
  The fatigue feelings of the patient will be assessed after each treatment, rated on a verbal analogue scale (VAS) ranging from 0 (no fatigue) to 10 (intolerable fatigue).

CONTACTS AND LOCATIONS:
Overall Officials: Georg Kranz, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No